CLINICAL TRIAL: NCT07343765
Title: Investigation of the Impact of Myomectomy on Uterine Artery Doppler Velocimetry Findings
Acronym: MYO-DOP
Status: Enrolling by invitation | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, İlke Esin Aydıner, M.D., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2025/276
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Leiomyoma (Uterine Fibroids); Myomectomy; Doppler Ultrasound
Keywords: leiomyoma; doppler; velocimetry; myomectomy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preoperative doppler measurements: Uterine leiomyoma cases before myomectomy operation will be investegated measuring doppler indices of pulsatility index, resistance index and systolic/dyastolic ratio.
- postoperative doppler measurements: Uterine leiomyoma cases who had myomectomy operation will be investegated measuring doppler indices of pulsatility index, resistance index and systolic/dyastolic ratio at the late postoperative period (40 days postoperatively)

SUMMARY:
Objective: This scientific study aims to investigate whether myomectomy induces significant changes in uterine artery blood flow patterns. While Doppler ultrasonography is traditionally used to assess myoma vascularity, differential diagnosis (adenomyoma or sarcoma), and fertility impacts, there is a lack of prospective evidence comparing preoperative and postoperative uterine artery Doppler findings.

Study Design and Rationale: The study will evaluate the hemodynamic influence of myomectomy by comparing flow measurements in the main uterine artery before and after surgical intervention. Existing literature has primarily focused on the correlation between myoma volume and vascular resistance; however, the direct impact of surgical removal of a myoma on uterine artery doppler velocimetry remains under-investigated.

Participant Involvement: Participation is entirely voluntary, and participants may withdraw at any time without any impact on their medical care. Data collection involves routine clinical history, physical examination, and non-invasive ultrasound measurements.

Clinical Significance: By establishing the effect of myoma removal on uterine blood supply, this research aims to provide guiding data for the follow-up and treatment planning of patients with leiomyomas. The findings may offer new insights into how surgical management restores or alters uterine hemodynamics, potentially influencing future diagnostic and therapeutic approaches.

DETAILED DESCRIPTION:
Uterine leiomyomas are the most common benign pelvic tumors in women and originate from the uterine smooth muscle tissue. While often asymptomatic, their size and location can cause clinical symptoms that significantly impair quality of life.

The pathogenesis of uterine leiomyoma is yet to be elucidated by the ongoing research. Our current knowledge reveals myoma pathogenesis involves a complex interplay of genetic factors, sex steroids, growth factors, extracellular matrix interactions, and angiogenesis. Understanding the mechanisms of leiomyoma pathogenesis and the interaction of myoma with adjacent myometrium is crucial to improve our management and treatment options.

Ultrasonography (USG) remains the gold standard for first-line imaging for uterine leiomyomas being highly sensitive, specific, and cost-effective. Doppler USG enables the evaluation of uterine blood flow by measuring the pulsatility index (PI), resistance index (RI), and systole/diastole (S/D) ratio. These parameters are widely used in routine obstetrics practice, where higher values indicate increased distal vascular resistance and lower values reflect enhanced perfusion and reduced impedance. Several studies observed increased blood flow in uterine artery measuring significantly lower resistance in the vessel. Our previous study revealed different doppler velocimetry findings in different leiomyoma localizations and a positive correlation between the indices and uterine operation history indicating an increased resistance in uterine artery after uterine surgery.

Myomectomy is a common procedure for cases of symptomatic leiomyoma and widely performed by gynecologists. This study aims to investigate the impact of myomectomy on uterine artery Doppler velocimetry parameters by comparing preoperative and postoperative measurements in patients diagnosed with uterine leiomyoma.

Method: This single-center, prospective clinical study will be conducted at the Bakırköy Dr. Sadi Konuk Training and Research Hospital, Department of Obstetrics and Gynecology, between August 2025 and January 2026. Following ethical approval, patients scheduled for myomectomy will be screened based on specific inclusion and exclusion criteria. Written informed consent will be obtained from all voluntary participants.

Patient data-including demographics, medical and obstetric history, presenting complaints (specifically abnormal uterine bleeding), and Visual Analog Scale (VAS) pain scores-will be recorded via the institutional electronic database (PROBEL). During routine gynecological assessment, transvaginal ultrasonography will be performed to determine myoma dimensions and localization according to the FIGO classification.

Uterine artery Doppler velocimetry findings, including the pulsatility index (PI), resistance index (RI), and systolic/diastolic (S/D) ratio, will be recorded both preoperatively and during the late postoperative period (after the 40th postoperative day). The histopathological findings will be integrated into the final analysis to confirm the diagnosis.

Statistical Analysis: Data analysis will be performed using SPSS Version 29.0.2 and G*Power 3.1.9.7.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged between 18 and 50 years.
* Women with uterine leiomyoma detected via ultrasonography.
* Patients referred to the Obstetrics and Gynecology department board for whom a myomectomy operation has been decided.
* Women who provide consent for transvaginal ultrasound examination.

Exclusion Criteria:

* Women under 18 years of age and postmenopausal women.
* Current pregnancy or postpartum status.
* Presence of known circulatory disorders, cardiovascular diseases, or other chronic conditions affecting blood flow.
* Smokers.
* Current use of hormonal medications (e.g., oral contraceptives, levonorgestrel-releasing intrauterine devices, etc.).
* Presence of concurrent gynecological pathologies (e.g., adenomyosis, endometriosis, ovarian cysts, or gynecological malignancies).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with uterus and uterine leiomyoma are enrolled.
Study Population: Patients scheduled for myomectomy at the Obstetrics and Gynecology Clinic of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pulsatility index | from the enrollment in preoperative period to the late postoperative period (40 days after operation)
  Pulsatility index will be measured in bilateral uterine arteries preoperatively and postoperatively in myomectomy cases.
resistance index | from the enrollment in preoperative period to the late postoperative period (40 days after operation)
  Uterine arter doppler measurement of resistance index will be measured preoperatively and postoperatively (40 days after operation) for bilateral uterine arteries.
systolic/dyastolic ratio | from the enrollment in preoperative period to the late postoperative period (40 days after operation
  Systolic/dyastolic ratio will be measured in bilateral uterine arteries preoperatively and postoperatively in myomectomy cases.

CONTACTS AND LOCATIONS:
Overall Officials: ilke esin aydıner, Principal Investigator — Bakırköy Sadi Konuk
Locations (1):
- Bakırköy Dr Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It has personal data of our participants and there is no consent of the participants regarding the sharing.

REFERENCES:
- [Background] Giuliani E, As-Sanie S, Marsh EE. Epidemiology and management of uterine fibroids. Int J Gynaecol Obstet. 2020 Apr;149(1):3-9. doi: 10.1002/ijgo.13102. Epub 2020 Feb 17. PMID 31960950
- [Background] Ciarmela P, Delli Carpini G, Greco S, Zannotti A, Montik N, Giannella L, Giuliani L, Grelloni C, Panfoli F, Paolucci M, Pierucci G, Ragno F, Pellegrino P, Petraglia F, Ciavattini A. Uterine fibroid vascularization: from morphological evidence to clinical implications. Reprod Biomed Online. 2022 Feb;44(2):281-294. doi: 10.1016/j.rbmo.2021.09.005. Epub 2021 Sep 20. PMID 34848152
- [Background] Stokes RE. Dangerousness and mental illness. Health Law Can. 1980 Summer;1(2):33, 39. No abstract available. PMID 10309430
- [Background] Drenhaus U, Dorka M. [Cause of tissue swelling during osmification following glutaraldehyde perfusion fixation]. Z Mikrosk Anat Forsch. 1985;99(1):146-60. No abstract available. German. PMID 3922145